CLINICAL TRIAL: NCT03168360
Title: Effect of Intensive Cognitive Rehabilitation in Subacute Stroke Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Yun-Hee Kim, MD, PhD, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-04-156
Record Dates: First submitted 2017-05-22; First posted 2017-05-30 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Stroke; Rehabilitation; Cognitive Function
MeSH Terms: conditions — Stroke | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive group (Experimental): cognitive rehabilitation therapy for 1 hour by cognitive therapist on every working day for 4 weeks
  Interventions: Procedure: Cognitive rehabilitation
- Conventional group (Active Comparator): cognitive rehabilitation therapy for 30 minutes by cognitive therapist on every working day for 4 weeks
  Interventions: Procedure: Cognitive rehabilitation

INTERVENTIONS:
Procedure: Cognitive rehabilitation — Intensive cognitive rehabilitation by cognitive therapist for 1 hours on every working day during subacute stroke phase

SUMMARY:
Early stroke rehabilitation is known to be an effective and essential therapy in gaining functional independence and preventing complications. However, there was no consensus of proper amount of cognitive rehabilitation in stroke patients. In this study, the investigators assess the effects of the intensive cognitive rehabilitation during subacute phase to improve cognitive function at 6 months after onset in patients with first-ever strokes.

DETAILED DESCRIPTION:
Intensive cognitive rehabilitation group

* cognitive therapy for 1 hours on every working day for 4 weeks

Conventional cognitive rehabilitation group

* cognitive therapy for 30 minutes on every working day for 4 weeks

ELIGIBILITY:
Inclusion Criteria:

* Acute first-ever stroke
* Korean Mini-Mental State Examination: 11~24 at 7 days after stroke onset

Exclusion Criteria:

* Transient ischemic stroke

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Korean-Montreal Cognitive Assessment (K-MoCA) | Change of K-MoCa after intensive cognitive rehabilitation for 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yun-Hee Kim, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chang WH, Sohn MK, Lee J, Kim DY, Lee SG, Shin YI, Oh GJ, Lee YS, Joo MC, Han EY, Kim YH. Korean Stroke Cohort for functioning and rehabilitation (KOSCO): study rationale and protocol of a multi-centre prospective cohort study. BMC Neurol. 2015 Mar 25;15:42. doi: 10.1186/s12883-015-0293-5. PMID 25886039
- [Derived] Clark B, Whitall J, Kwakkel G, Mehrholz J, Ewings S, Burridge J. The effect of time spent in rehabilitation on activity limitation and impairment after stroke. Cochrane Database Syst Rev. 2021 Oct 25;10(10):CD012612. doi: 10.1002/14651858.CD012612.pub2. PMID 34695300
- [Derived] Longley V, Hazelton C, Heal C, Pollock A, Woodward-Nutt K, Mitchell C, Pobric G, Vail A, Bowen A. Non-pharmacological interventions for spatial neglect or inattention following stroke and other non-progressive brain injury. Cochrane Database Syst Rev. 2021 Jul 1;7(7):CD003586. doi: 10.1002/14651858.CD003586.pub4. PMID 34196963